CLINICAL TRIAL: NCT01794312
Title: Efficacy and Safety Assessment of T4020 Versus Vehicule in Patients With Chronic Neurotrophic Keratitis or Corneal Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LT4020-PIII-12/11
Record Dates: First submitted 2013-01-25; First posted 2013-02-18 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Keratitis; Corneal Ulcer
MeSH Terms: conditions — Keratitis; Corneal Ulcer | interventions — Pharmaceutical Vehicles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T4020 (Experimental): One drop every 2 days
  Interventions: Device: T4020
- Vehicle (Placebo Comparator): One drop every 2 days
  Interventions: Device: Vehicle

INTERVENTIONS:
Device: T4020
  Arms: T4020
Device: Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to assess the efficacy and safety of T4020 versus vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with one chronic keratitis/corneal ulcer
* Patients who signed and dated informed consent

Exclusion Criteria:

* Patient under 18 years
* Patient with a perforated corneal ulcer OR any risk of immediate perforation of corneal ulcer.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Development Director, Clermont-Ferrand, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T4020 | Vehicle
Started | 74 | 78
Completed | 68 | 67
Not Completed | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T4020 | Vehicle | Total
Number analyzed (Participants) | 74 | 78 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 37 | 32 | 69
  >=65 years | 37 | 45 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (17) | 65.2 (17.8) | 63.8 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 34 | 36 | 70
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 16 | 20 | 36
  Poland | 12 | 14 | 26
  Turkey | 8 | 7 | 15
  Belgium | 6 | 8 | 14
  Italy | 7 | 6 | 13
  Spain | 7 | 5 | 12
  Greece | 6 | 6 | 12
  Switzerland | 4 | 4 | 8
  Netherlands | 4 | 4 | 8
  Sweden | 2 | 1 | 3
  United Kingdom | 1 | 2 | 3
  Austria | 0 | 1 | 1
  Portugal | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction in Neurotrophic the Keratitis/Ulcer Area on Day28
Description: Reduction in neurotrophic ulcer/keratitis area of 50% or more
Time Frame: Day 28
Population: Modified Intent to treat (m-ITT): All randomised patients received at least 1 IMP dose, with at least 1 baseline and 1 post-baseline efficacy assessment.
  For the primary outcome measure, 4 patients (2 in the T4020 and Vehicle groups) had no data for the reduction from baseline of corneal ulcer/keratitis area and were not included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | T4020 | Vehicle
Number analyzed (Participants) | 72 | 76
Participants | 37 | 44

2. Secondary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event
Description: With at least one TEAE
Time Frame: From the first visit to the final visit performed by the patient + 1 month later, assessed up to 71 days
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | T4020 | Vehicle
Number analyzed (Participants) | 74 | 78
Participants | 25 | 27

3. Secondary Outcome: Best Corrected Visual Acuity
Description: Change from baseline in far best-corrected visual acuity (LogMAR) in the pathologic eye
Time Frame: Baseline and Day 28
Population: Safety set
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | T4020 | Vehicle
Number analyzed (Participants) | 74 | 78
LogMAR | -0.055 (0.362) | -0.035 (0.590)

ADVERSE EVENTS:
Time Frame: From the first visit to the final visit performed by the patient + 1 month later, assessed up to 71 days
Groups:
- T4020; Vehicle: One drop 4 times per week
Arm/Group | T4020 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/78
Serious Adverse Events (participants affected / at risk) | 3/74 | 7/78
Other Adverse Events (participants affected / at risk) | 25/74 | 27/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T4020 (N=74) | Vehicle (N=78)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Herpes Simplex ophthalmic (Infections and infestations) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Corneal neovascularisation (Eye disorders) | 0 (0) | 1 (1)
Corneal infection (Infections and infestations) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Corneal perforation (Eye disorders) | 0 (0) | 1 (1)
Keratitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T4020 (N=74) | Vehicle (N=78)
Ulcerative keratitis (Eye disorders) | 3 (3) | 4 (4) — Ocular adverse event in pathologic eye
Hypopyon, Keratitis bacterial, Keratitis herpetic, Corneal infection, Dacryocanaliculitis, Dacryocys (Infections and infestations) | 3 (3) | 9 (9) — Ocular adverse event in pathologic eye
Instillation site reaction (General disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Vital dye staining cornea present (Investigations) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Hyperaemia (Vascular disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Conjuncticitis allergic, diplopia (Eye disorders) | 1 (1) | 1 (1) — Ocular adverse event in the other eye
Device related infection, Gastroenteritis, Oral herpes, Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0) — Non ocular adverse event
Headache (Nervous system disorders) | 0 (0) | 3 (3) — Non ocular adverse event
Femoral neck fracture, Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Non ocular adverse event
Influenza like illness (General disorders) | 0 (0) | 1 (1) — Non ocular adverse event
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) — Non ocular adverse event
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Non ocular adverse event
Begnin prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Non ocular adverse event
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Non ocular adverse event
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) — Non ocular adverse event
Keratitis (Eye disorders) | 3 (3) | 1 (1) — Ocular adverse event in pathologic eye
Eye pain (Eye disorders) | 0 (0) | 3 (3) — Ocular adverse event in pathologic eye
Eye irritation (Eye disorders) | 2 (2) | 0 (0) — Ocular adverse event in pathologic eye
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event in pathologic eye
Acanthamoeba keratitis (Eye disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Conjunctival hemorrhage (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event in pathologic eye
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event in pathologic eye
Corneal epithelium defect (Eye disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Corneal erosion (Eye disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Corneal neovascularisation (Eye disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Corneal perforation (Eye disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Diplopia (Eye disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Dry eye (Eye disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event in pathologic eye
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event in pathologic eye
Neurotrophic keratopathy (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event in pathologic eye
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Punctate keratitis (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event in pathologic eye
Uveitis (Eye disorders) | 0 (0) | 1 (1) — Ocular adverse event in pathologic eye
Vision blurred (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event in pathologic eye
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event in pathologic eye
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event in pathologic eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever form without prior written agreement of THEA.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT01794312/Prot_SAP_000.pdf